CLINICAL TRIAL: NCT01568281
Title: A Randomised, Open Label, Single Centre, 2 Way Crossover Bioequivalence Study Comparing Arimidex Tablet 1 mg and Anastrozole Orally Rapid Disintegration Film Formula 1 mg After Single Oral Administration in Japanese Healthy Male Subjects
Brief Title: Bioequivalence Study Comparing Arimidex Tablet and Anastrozole ODF in Japanese Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D539EC00001
Record Dates: First submitted 2012-03-28; First posted 2012-04-02 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-06

CONDITIONS: Safety; Pharmacokinetics
Keywords: Bioequivalence; pharmacokinetics; safety; anastrozole; Arimidex; Japanese; healthy subject
MeSH Terms: interventions — Anastrozole

ARMS (4):
- 1 (Experimental): 2 way crossover
  Interventions: Drug: Anastrozole ODF
- 2 (Experimental): 2 way crossover
  Interventions: Drug: Arimidex tablet
- 3 (Experimental): 2 way crossover
  Interventions: Drug: Anastrozole ODF
- 4 (Experimental): 2 way crossover
  Interventions: Drug: Arimidex tablet

INTERVENTIONS:
Drug: Anastrozole ODF — Each volunteer will receive a single dose of Anastrozole ODF with water.
  Arms: 1
Drug: Arimidex tablet — Each volunteer will receive a single dose of Arimidex tablet with water
  Arms: 2
Drug: Anastrozole ODF — Each volunteer will receive a single dose of Anastrozole ODF without water.
  Arms: 3
Drug: Arimidex tablet — Each volunteer will receive a single dose of Arimidex tablet with water
  Arms: 4

SUMMARY:
This study is to investigate whether anastrozole ODF is bioequivalent with Arimidex tablet after a single oral administration of each anastrozole formulation.

DETAILED DESCRIPTION:
A Randomised, Open label, Single centre, 2 way Crossover Bioequivalence Study Comparing Arimidex Tablet 1 mg and Anastrozole Orally Rapid Disintegration Film Formula 1 mg After Single Oral Administration in Japanese Healthy Male Subjects

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures Japanese healthy male subjects aged 20 to 45 years Male subjects should be willing to use barrier contraception ie, condoms, until 3 months after the last dose of investigational product Have a body mass index (BMI) between 18 and 27 kg/m2

Exclusion Criteria:

* History of any clinically significant disease or disorder
* History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs Any clinically significant illness, medical/surgical procedure or trauma
* Any clinically significant abnormalities in clinical chemistry, haematology or urinalysis results

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2012-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Investigation whether anastrozole ODF is bioequivalent with Arimidex tablet. | Blood samples are taken repeatedly for 24 hours and also taken occasionally up to 168 hours after each dose
  By assessment of AUC and Cmax of anastrozole after a single oral administration of each anastrozole formulation.

SECONDARY OUTCOMES:
Evaluation of the pharmacokinetic properties of Arimidex tablet and anastrozole ODF following a single oral dose. | Blood samples are taken repeatedly for 24 hours and also taken occasionally up to 168 hours after each dose
  By assessment of AUC, MRT, tmax, kel and t1/2 of anastrozole.
Evaluation of the safety and tolerability of Anastrozole ODF 1 mg. | Safety variables are measured prior to treatment and up to 14 to 17 days (follow-up) after the last dose. Subjects will be monitored throughout the study for adverse events
  By assessment of adverse events, clinical laboratory tests, 12-lead ECG, blood pressure, pulse rate and body temperature.

CONTACTS AND LOCATIONS:
Overall Officials: Eisei Shin, MD, Study Director — AstraZeneca R&D Japan; Kyoko Matsuguma, MD PhD, Principal Investigator — Kyushu Clinical Pharmacology Research Clinic
Locations (1):
- Research Site, Fukuoka, Fukuoka, Japan